CLINICAL TRIAL: NCT06669468
Title: Comparison of the Efficacy of Perineal and Anal Electrical Stimulation in Patients with Urinary Incontinence After Radical Prostatectomy. a Prospective Randomised Controlled Trial
Brief Title: Comparison of the Efficacy of Perineal and Anal Electrical Stimulation in Patients with Urinary Incontinence After Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PamukkaleU.ftr-NYıldız-002
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Prostatectomy; Urinary Incontinence
Keywords: Anal Electrical Stimulation; Perineal Electrical Stimulation; Radical Prostatectomy; İncontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — pentalenolactone F methyl ester

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: PFME (Active Comparator): The patients were instructed to do as an home exercise program in first 2 weeks, 5 s contraction and 10 s relaxation, including two sets of 5 repetition daily, in following 2 weeks 10 s contraction and 20 s relaxation, including two sets of 10 repetition daily, and after 4 weeks, 10 s contraction and 20 s relaxation including three sets of 10 repetition daily in three different position (lying, sitting, and standing). So in the first 2 weeks 30 contractions daily, in following 2 weeks 60 contractions daily and upward 4th weeks, 90 contractions daily with progressively increasing intensity was done. All patients were asked to mark the exercise at a daily home schedule. Patients who did not complete more than 20% of the list according to the daily home program were excluded from the study.
  Interventions: Other: PFME
- Group 2: PFME + Anal ES (Experimental): Anal ES was applied in the lithotomy position by means of a combined electrotherapy (stimulation) device with anal electrodes. Anal ES was applied 3 days a week, 20 minutes a day, for a total of 24 sessions for 8 weeks. Stimulation parameters were 50 Hz frequency, 5-10 s work-rest cycle and 300 µs pulse amplitude. Symmetrical biphasic pulse wave was given in the range of 1-100 mA (according to the patient's discomfort level feedback). In this procedure, it was applied with an anal probe placed in the anal region. Patients did not perform voluntary contractions during ES. Anal probes were used separately for each patient. Anal ES sessions were performed by an investigator participating in the study. Men who missed any treatment session for the stimulation group were excluded from the study.
  Interventions: Other: PFME + Anal ES
- Group 3: PFME + Perineal ES (Experimental): Perineal ES was applied in the lithotomy position by means of a combined electrotherapy (stimulation) device with surface electrodes. Anal ES was applied 3 days a week, 20 minutes a day, for a total of 24 sessions for 8 weeks. Stimulation parameters were 50 Hz frequency, 5-10 s work-rest cycle and 300 µs pulse amplitude. Symmetrical biphasic pulse wave was given in the range of 1-100 mA (according to the patient's discomfort level feedback). In this procedure, five surface electrodes with a diameter of 2 cm will be used, four electrodes symmetrically in the perianal region and one electrode in the leg (ground-neutral electrode). Patients will not perform voluntary contractions during ES. Surface electrodes will be used separately for each patient. Perineal ES sessions were performed by an investigator participating in the study. Men who missed any treatment session for the stimulation group were excluded from the study.
  Interventions: Other: PFME + Perineal ES

INTERVENTIONS:
Other: PFME — All patients were asked to mark the exercise at a daily home schedule. Patients who did not complete more than 20% of the list according to the daily home program were excluded from the study.
  Arms: Group 1: PFME
Other: PFME + Anal ES — Anal ES was applied 3 days a week, 20 minutes a day, for a total of 24 sessions for 8 weeks.
  Arms: Group 2: PFME + Anal ES
Other: PFME + Perineal ES — Perineal ES was applied 3 days a week, 20 minutes a day, for a total of 24 sessions for 8 weeks.
  Arms: Group 3: PFME + Perineal ES

SUMMARY:
Radical prostatectomy (RP) is a common procedure for the treatment of prostate cancer. However, postoperative urinary incontinence (UI) is an important reason for morbidity. UI negatively affects the quality of life in 30-50% of patients, especially in the early period (3 weeks to 6 months). However, it takes approximately 1 year to achieve continence (1).

Conservative treatment methods include pelvic floor muscle exercises (PFME) with or without biofeedback (BF), anal and perineal electrical stimulation (ES), magnetic stimulation (MS), compression (penile clamps), lifestyle changes and combinations of these methods (2).

ES artificially stimulates the pudendal nerve and its branches to cause direct and reflex responses of the urethral and periurethral striated muscles in women. ES also inhibits detrusor overactivity (3,4). There is conflicting evidence as to whether the addition of ES to treatment increases the efficacy of PFME alone in patients with UI after RP (Level of evidence:1b), (5). However, ES may benefit PFME for up to six months (Level of evidence: 2b), (5). Non-neurogenic male incontinence guidelines recommend PFME alone or in combination with BF and/or ES for men undergoing RP to accelerate improvement of UI (5).

Many studies have shown that anal ES alone (1,7,8) or in combination with PFME (4,9,10,11) is more effective than untreated (4,7,9,11) or placebo ES (8,12). There are only two randomised controlled trials in the literature evaluating the efficacy of perineal ES in patients with UI after RP (13,14). In the study by Yıldız et al. (13), the group receiving perineal ES and the control group receiving no treatment were compared in patients who developed UI after RP. The results showed that incontinence severity, incontinence episodes, quality of life and anxiety parameters improved significantly in the 8th week in the group receiving perineal ES compared to the control group. In the study by Pané-Alemany et al. (14), a group receiving perianal ES and a group receiving anal ES were compared in patients who developed UI after RP. In the study, it was shown that the efficacy of the two treatments was not statistically different.

Our study is the first prospective randomised controlled trial to evaluate the efficacy of perineal and anal ES added to PFME in patients with UI after RP. The aim of this study was to evaluate the efficacy of perineal ES and anal ES added to PFME on clinical parameters related to UI, quality of life and sexual functions, depression and anxiety. In addition, patients' preparation time for stimulation, treatment satisfaction and discomfort levels will be evaluated.

DETAILED DESCRIPTION:
The research will be conducted at Pamukkale University Physical Medicine and Rehabilitation (PMR) Department, Urogynecological Rehabilitation Unit between November 2024 and January 2025.

The study included 93 patients (described in detail in the statistics section) who accepted the treatment among the male patients who applied to Pamukkale University FTR Polyclinic with the complaint of UI after RP or who were referred to the Urogynecological Rehabilitation Unit by the Urology outpatient clinic and who met the inclusion criteria. Patients will be informed about the content, purpose and application of the study and their written consent will be obtained.

At the beginning of the study, age, height, weight, education level, occupation, marital status, previous operations, systemic diseases, alcohol, tea, coffee, coffee, cigarette use and medications will be questioned in patients who applied to Pamukkale University FTR Polyclinic or Urology Polyclinic with the complaint of UI after RP and referred to the Urogynecological Rehabilitation Unit. The type of UI (stress, urge, mixed, drip) will be determined in all patients participating in the study.

Patients will be advised to continue their medical treatments for reasons other than incontinence during the treatment period. No lifestyle modification recommendations regarding urinary function will be given during the treatment period and participants will be instructed not to change their habits during the 8-week period of the study.

Ninety-three male patients who meet the inclusion and exclusion criteria after RP will be randomly divided into three groups using a random number table. The first group will receive PFME, the second group will receive PFME + anal ES, and the third group will receive PFME + perineal ES.

Group 1: PFME Group 2: PFME + anal ES Group 3: PFME + perineal ES

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Men with RP with incontinence over >50 g/24 h and no residual cancer after RP on pathological examination
* Men within 1 month to 1 year after catheter removal
* Willingness to complete and do the QoL scale.
* Understanding procedures, benefits, and possible side effects.
* Being able to give written, informed consent.

Exclusion Criteria:

* UI history before RP.
* History of conservative treatment after RP including ES.
* Prolonged indwelling urethral catheterization (more than 15 days).
* Previous urological surgery history.
* Men receiving radiotherapy.
* Presence of urethral stricture and urinary tract infection.
* Heart failure, presence of a pacemaker, implanted defibrillator.
* Transurethral resection of the prostate due to benign prostatic hyperplasia.
* Use of drugs that may affect bladder function (antimuscarinic, duloxetine, tricyclic antidepressant, etc.).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 93 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Severity of incontinence | 8 weeks
  The 24-hour pad test was carried out to evaluate urinary loss.

SECONDARY OUTCOMES:
Incontinence episodes | 8 weeks
  Patients with a 50% or greater reduction in incontinence episodes were consider improvement
Three-day Bladder Diary | 8 weeks
  It was used "frequency of voiding", "incontinence episodes", "nocturia", "number of pads" from data collected with a 3-day bladder diary.
Quality of Life - Incontinence Impact Questionnaire (IIQ-7) | 8 weeks
  The IIQ-7 scale which has great validity in studies was used to assess the patient's QoL associated with incontinence problem
Level of sexual function - International Index of Erectile Function (IIEF) | 6 weeks
  Sexual functions
Level of Anxiety and Depression - Hospital Anxiety and Depression Scale (HAD) | 8 weeks
  Anxiety and Depression
Treatment satisfaction - Likert scale (1-5 ) | 8 weeks
  The patients evaluated the change of their urinary incontinence on a 5-point Likert scale (5, very satisfied; 4, satisfied; 3, equally satisfied and unsatisfied; 2, unsatisfied; 1, very unsatisfied)
Treatment Success (Continence rate) | 8 weeks
  Patients with ≤8 gr in 24-hour pad test measurement will be considered "continent"
Cure (Dry) and Improvement Rate | 8 weeks
  the absence of will be evaluated as "dryness"

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin YILDIZ Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No